CLINICAL TRIAL: NCT07249749
Title: Factors Associated With Mortality in the Intensive Care Unit From the Orinoco Region. An Observational Trial
Brief Title: Factor Associated With Mortality in the ICU
Acronym: ICUMortal
Status: Not yet recruiting | Type: Observational
Sponsor: Hospital Departamental de Villavicencio (Other)
Responsible Party: Principal Investigator, Norton Perez-Gutierrez, MD, ICU director, Hospital Departamental de Villavicencio
Other Study IDs: GRIVI_2025_02_UCI_MORTAL
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Critically Ill; Intensive Care (ICU); Intensive Care Medicine; Mortality; Mortality Prediction; Mortality in Intensive Care Units
Keywords: Critically Ill; Intensive Care Unit; Mortality; Colombia
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ICU mortality: Patients who died in the intensive care unit within the first 28 days of admission.
  Interventions: Other: Exposure factors
- ICU survivors: Patients discharged from the intensive care unit alive within the first 24 days.
  Interventions: Other: Exposure factors

INTERVENTIONS:
Other: Exposure factors — Evaluation of factors associated with mortality

SUMMARY:
ICU mortality indicates the severity of disease, healthcare quality, and the efficacy of interventions. The severity scores are tools to predict the risk of mortality in the ICU, and the APACHE II score is frequently used for this purpose. However, studies validating the score in Colombia are limited. There is uncertainty about the precision and discrimination capacity of the APACHE II score in a population that varies from the original, with varying diseases, and in a different timeline. The investigators determined to evaluate: 1. Evaluate the rate of mortality in the ICU by type of disease and type of admission. 2. The factors associated with mortality. 3. Validate the performance of the APACHE II score as a predictor of mortality.

DETAILED DESCRIPTION:
Introduction Mortality serves as an indicator of healthcare quality in the intensive care unit. The APACHE II score is a practical tool for predicting mortality, though its application varies. Studies validating the APACHE II score in Colombia are limited. This study aimed to evaluate the performance of the Acute Physiology and Chronic Health Evaluation (APACHE) II score as a predictor of mortality in the intensive care unit of a hospital in Villavicencio, Colombia.

Methodology Design: In this single-center, retrospective cohort, consecutive cases were observed from admission to discharge from the ICU. The demographic characteristics, diagnosis type, admission origin, and APACHE II score were systematically calculated on a database, and the cases were divided into two populations for comparison based on the outcome.

Setting: The study was performed in the ICU of Hospital Departamental de Villavicencio, a reference institution for the Orinoco region. It has 350 beds, four adult polyvalent critical care units with 40 beds, and the only oncology unit in the zone.

Patients: Critically ill patients admitted from January 2022 to June 2025 were included.

Sample: The study included all patients in the discharge database and used no sampling method.

Inclusions: All adult patients older than 18 years admitted during the study period were included.

Exclusions: The analysis excluded patients admitted as intermediate care (low therapeutic intervention with a TISS [Therapeutic Intervention Scoring System]-28 score below 20 points).

Data collection: The information of all patients admitted to the ICU was systematically collected from the clinical chart on discharge and uploaded to an electronic database in a standardized online format. The severity score was calculated within the first 24 hours of admission. Demographic characteristics, insurance, diagnosis information, APACHE II score, TISS-28 score, mechanical ventilation duration, and outcome were recorded. The outcomes evaluated were mortality (early or late), ICU length of stay, and mechanical ventilation duration.

Analysis plan: The investigators used Jamovi 2.6.44 program for the analysis, and Prism 10.6.1 or Wizard 1.9.49 for the graphics. Categorical variables are presented as frequencies and proportions; continuous variables are presented as their central tendency and dispersion, after verifying normality. The Chi-square test was selected to compare categorical variables, and the t-test or the Mann-Whitney test to compare quantitative variables. A value of p < 0.01 was chosen as statistical significance. A logistic regression analysis was performed to confirm the effect of APACHE II score on the outcome. Observed mortality rate (early or late [more than 48 hours) was compared with the expected rate (standardized or SMR). The discrimination of the score was determined by the area under the curve (AUC) of the receiver operating characteristic (ROC), with a closer value to 1 for diagnosis and type of admission.

Ethical aspects: The hospital research committee previously approved the database analysis and waived informed consent, as the study was classified as low-risk research in accordance with national regulations. The project was registered on the platform ClinicalTrials.gov in accordance with the Helsinki Declaration, including observational trials.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients older than 18 admitted to the intensive care unit during the study period.

Exclusion Criteria:

* Patients admitted for intermediate care (low therapeutic intervention with a TISS [Therapeutic Intervention Scoring System] - 28 score below 20 points). Patients derived to other institutions.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult critically ill patients with a high need of support and intervention in the intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2028-12-20 (Estimated); Study Completion 2028-12-21 (Estimated)

PRIMARY OUTCOMES:
Mortality | Within 28 days
  Dead discharges

CONTACTS AND LOCATIONS:
Overall Officials: Norton Perez Gutierrez, MD, Principal Investigator — Hospital Departamental de Villavicencio
Locations (1):
- Hospital Departamental de Villavicencio, Villavicencio, Meta Department, Colombia

IPD SHARING:
Plan to Share IPD: No
The data contains sensitive information from patients.

REFERENCES:
- [Result] Sudarsanan S, Sivadasan P, Chandra P, Omar AS, Gaviola Atuel KL, Ulla Lone H, Ragab HO, Ehsan I, Carr CS, Pattath AR, Alkhulaifi AM, Shouman Y, Almulla A. Comparison of Four Intensive Care Scores in Predicting Outcomes After Venoarterial Extracorporeal Membrane Oxygenation: A Single-center Retrospective Study. J Cardiothorac Vasc Anesth. 2025 Jan;39(1):131-142. doi: 10.1053/j.jvca.2024.10.027. Epub 2024 Oct 22. PMID 39550342
- [Result] Li X, Yi Q, Luo Y, Wei H, Ge H, Liu H, Zhang J, Li X, Xie X, Pan P, Zhou H, Liu L, Zhou C, Zhang J, Peng L, Pu J, Yuan J, Chen X, Tang Y, Zhou H. Prediction Model of In-Hospital Death for Acute Exacerbation of Chronic Obstructive Pulmonary Disease Patients Admitted to Intensive Care Unit: The PD-ICU Score. Respiration. 2025;104(2):85-99. doi: 10.1159/000541367. Epub 2024 Sep 11. PMID 39260355
- [Result] Knaus WA, Zimmerman JE, Wagner DP, Draper EA, Lawrence DE. APACHE-acute physiology and chronic health evaluation: a physiologically based classification system. Crit Care Med. 1981 Aug;9(8):591-7. doi: 10.1097/00003246-198108000-00008. PMID 7261642
- [Result] Chlabicz M, Laguna W, Kazimierczyk R, Kazimierczyk E, Lopatowska P, Gil M, Sobkowicz B, Kaminski KA, Tycinska A. Value of APACHE II, SOFA and CardShock scoring as predictive tools for cardiogenic shock: A single-centre pilot study. ESC Heart Fail. 2024 Dec;11(6):3584-3597. doi: 10.1002/ehf2.15020. Epub 2024 Aug 13. PMID 39136422
- [Result] Liengswangwong W, Siriwannabhorn R, Leela-Amornsin S, Yuksen C, Sanguanwit P, Duangsri C, Kusonkhum N, Saelim P. Comparison of Modified Early Warning Score (MEWS), Simplified Acute Physiology Score II (SAPS II), Sequential Organ Failure Assessment (SOFA), and Acute Physiology and Chronic Health Evaluation II (APACHE II) for early prediction of septic shock in diabetic patients in Emergency Departments. BMC Emerg Med. 2024 Sep 4;24(1):161. doi: 10.1186/s12873-024-01078-8. PMID 39232644
- [Result] Tekin B, Kilic J, Taskin G, Solmaz I, Tezel O, Basgoz BB. The Comparison of scoring systems: SOFA, APACHE-II, LODS, MODS, and SAPS-II in critically ill elderly sepsis patients. J Infect Dev Ctries. 2024 Jan 31;18(1):122-130. doi: 10.3855/jidc.18526. PMID 38377099